CLINICAL TRIAL: NCT06254612
Title: A Multi-center, Double-Blind, Randomized, Placebo-Controlled Study of the Efficacy and Safety of SP-624 in the Treatment of Adults With Major Depressive Disorder
Brief Title: A Study of the Efficacy and Safety of SP-624 in the Treatment of Adults With Major Depressive Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sirtsei Pharmaceuticals, Inc. (Industry)
Collaborators: Rho, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP-624-202
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SP-624 (Experimental): Participants to receive two 10 mg capsules of SP-624 once daily for a total daily dose of 20 mg
  Interventions: Drug: SP-624
- Placebo (Placebo Comparator): Participant to receive 2 matching placebo capsules once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SP-624 — Once daily oral administration of two capsules totaling 20 mg/day
  Arms: SP-624
Drug: Placebo — Once daily oral administration of two matching placebo capsules
  Arms: Placebo

SUMMARY:
This is a Phase 2B clinical study evaluating the effectiveness and safety of SP-624 as compared to placebo in the treatment of adults with Major Depressive Disorder.

ELIGIBILITY:
Key Inclusion Criteria:

* Males and females, aged 18 to 65 years, inclusive.
* Meet DSM-5 criteria for moderate to severe MDD, as confirmed by the Mini International Neuropsychiatric Interview (MINI).
* In generally good physical health, in the opinion of the Investigator.
* Body mass index (BMI) must be ≥ 18 and ≤ 45 kg/m2.

Key Exclusion Criteria:

* Female who is pregnant, breastfeeding, or less than 6 months postpartum at screen.
* A history of or current DSM-5 diagnosis of MDD with psychotic features, any schizophrenia spectrum and other psychotic disorders, bipolar disorder, or personality disorder.
* Presence or history of any known clinically significant cardiovascular disorders including, but not limited to: coronary artery disease, heart failure, valvular heart disease, cardiomyopathies, myocardial infarction, chamber enlargement or hypertrophy, or orthostatic hypotension.
* Presence of uncontrolled hypertension, defined as consistent sitting systolic blood pressure (SBP) >160 mmHg or consistent sitting diastolic blood pressure (DBP) >95 mmHg despite present therapy.
* Screening laboratory value(s) outside the laboratory reference range that are considered to be clinically significant by the Investigator (clinical chemistry, hematology, thyroid function, and urinalysis).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Montgomery-Asberg Depression Rating Scale (MADRS) total score. | Baseline to Week 4
  The MADRS is a 10-item depression rating scale used to assess the severity of depression. Individual items are scored on a 7-point scale (0 to 6). The toal score is the sum of individual items, ranging from 0 to 60; where a higher score indicates more depression.

SECONDARY OUTCOMES:
Change from Baseline in the Clinical Global Impression - Severity (CGI-S) score. | Baseline to Weeks 1-4 and 1- and 2- Week Follow-up
  The CGI-S is a 7-point scale to rate the severity of the participant's illness at the time of assessment, relative to the clinician's past experience with participants who have the same diagnosis. A score of 1 represents "normal" and 7 represents "most extremely ill".
Change from Baseline in Quick Inventory of Depressive Symptomology-Self-Report (QIDS-SR) total score. | Baseline to Weeks 1-4 and 1- and 2- Week Follow-up
  The QIDS-SR is a 16-item self-reported scale where each item has a 4-point scale where 0 represents least impact scores while 3 represents greatest impact scores. Some questions are linked. The total score ranges from 0 to 27 where a higher score indicates more depression.
Change from Baseline in the Montgomery-Asberg Depression Rating Scale (MADRS) total score. | Baseline to Weeks 1-3 and 1- and 2- Week Follow-up
  The MADRS is a 10-item depression rating scale used to assess the severity of depression. Individual items are scored on a 7-point scale (0 to 6). The toal score is the sum of individual items, ranging from 0 to 60; where a higher score indicates more depression.
Change from Baseline in 17-item-Hamilton Depression Rating Scale (HAM-D-17) total score. | Baseline to Weeks 2 and 4
  The 17-item HAM-D is used to assess the severity of depression. Individual items are scored on either a 3-point (0 to 2) or a 5-point scale (0 to 4), with 0=No difficulty/absent and 4=most severe. The total score is the sum of individual items, ranging from 0 to 52; where a higher score indicates more depression.
Change from Baseline in Sheehan Disability Scale (SDS) total score. | Baseline to Weeks 2 and 4
  The SDS is a 3-part scale that measures the degree of disruption on work, social and family life using an 11-point scale where 0 represents "no disruption" and 10 represents "extreme disruption". In addition to the 11-point scale, participants are asked to indicate the number of days in the past week that were "lost" and numbers of days that were "underproductive". The results of these questions have a range from 0 to 7. A total global functioning impairment score can be utilized by summing the scores from work, social and family life scales for a value range from 0 to 30.
Change from Baseline in Symbol Digit Modalities Test (SDMT) score. | Baseline to Weeks 2 and 4
  The SDMT is an assessment of complex scanning and visual tracking requiring elements of attention, visuoperceptual processing, working memory, and cognitive/psychomotor speed. The SDMT measures the time to pair abstract symbols with specific numbers. The number of correct substitutions within 90 seconds is recorded and the total score is derived from the total number of correct responses with a minimum possible score of 0 and maximum of 110 where high scores indicate better outcome.
Incidence rates of treatment emergent adverse events (TEAEs), serious adverse events (SAEs), and TEAEs leading to withdrawal from study. | Baseline to Weeks 1-4 and 1- and 2- Week Follow up

CONTACTS AND LOCATIONS:
Overall Officials: Greg Rigdon, PhD, Study Director — Sirtsei Pharmaceuticals, Inc.
Locations (50):
- United States (50):
  - IMA Clinical Research, Phoenix, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - SanRo Clinical Research Group, Bryant, Arkansas
  - Clinical Innovations, Bellflower, California
  - Sun Valley Research Center, Imperial, California
  - Sunwise Clinical Research, Lafayette, California
  - Synergy San Diego, Lemon Grove, California
  - Excell Research, Oceanside, California
  - CiTrials, Riverside, California
  - Collaborative Neuroscience Research, Torrance, California
  - Next Level Clinical Trials, West Covina, California
  - MCB Clinical Research Centers, Colorado Springs, Colorado
  - Clinical Neuroscience Solutions, Jacksonville, Florida
  - Accel Clinical, Lakeland, Florida
  - Segal Trials, Lauderhill, Florida
  - Segal Trials - Miami Lakes, Miami Lakes, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - DMI Research, Pinellas Park, Florida
  - Accelerated Enrollment Solutions, Atlanta, Georgia
  - Velocity Clinical Research, Meridian, Idaho
  - Revive Research Institute, Elgin, Illinois
  - Tandem Clinical Research, Marrero, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - Neurobehavioral Medicine Group, Bloomfield Hills, Michigan
  - Midwest Research Group, Saint Charles, Missouri
  - Alivation Research, Lincoln, Nebraska
  - IMA Clinical Research, Las Vegas, Nevada
  - Redbird Research, Las Vegas, Nevada
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - CenExel HRI, Marlton, New Jersey
  - IMA Clinical Research, Albuquerque, New Mexico
  - Integrative Clinical Trials, Brooklyn, New York
  - Pioneer Clinical Research, New York, New York
  - Magnolia Clinical Research, Cary, North Carolina
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - New Hope Clinical Research, Charlotte, North Carolina
  - Velocity Clinical Research, Beachwood, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - North Star Medical Research, Middleburg Heights, Ohio
  - Summit Headlands, Portland, Oregon
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Clinical Neuroscience Solutions, Memphis, Tennessee
  - Donald J. Garcia, Jr, MD, PA, Austin, Texas
  - Future Search Trials of Dallas, Dallas, Texas
  - Haracec Clinical Research, El Paso, Texas
  - Pillar Clinical Research, Richardson, Texas
  - R and H Clinical Research, Stafford, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
  - Core Clinical Research, Everett, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raskin J, Clayton AH, Kornstein SG, Papakostas GI, Prescott Y, Abernathy K, Hall J, Ackermann M, Wargin W, Rigdon G; SP-624-201 study investigators. A phase 2, multicenter, double-blind, randomized, placebo-controlled study of the safety and efficacy of forvisirvat (SP-624) in the treatment of adults with major depressive disorder. Curr Med Res Opin. 2025 Sep;41(9):1723-1734. doi: 10.1080/03007995.2025.2574465. Epub 2025 Oct 29. PMID 41099447